CLINICAL TRIAL: NCT01112839
Title: Reducing Breast Cancer Recurrence With Weight Loss: A Vanguard Trial
Brief Title: Reducing Breast Cancer Recurrence With Weight Loss
Acronym: ENERGY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Washington University School of Medicine (Other); University of Colorado, Denver (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Cheryl Rock, Study Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CA148791-01
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer; Overweight; Obesity
Keywords: Overweight; Obese; Breast cancer survivors; Weight loss; Exercise; Physical activity
MeSH Terms: conditions — Breast Neoplasms; Overweight; Obesity; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Less Intensive Group (Active Comparator): Participants in this group would receive print materials on diet and exercise and two individual counseling sessions; one at the beginning of the study and another 6 months later.
  Interventions: Behavioral: Less Intensive
- Intensive Group (Experimental): Participants in this group would receive print materials on diet and exercise and attend group sessions that would meet weekly for the first 4 months, then every two weeks for the next 2 months, and then monthly for the next 6 months over the course of one year.
  Interventions: Behavioral: Intensive Group

INTERVENTIONS:
Behavioral: Less Intensive — Participants in this group would receive print materials on diet and exercise and two individual counseling sessions; one at the beginning of the study and another 6 months later.
  Arms: Less Intensive Group
Behavioral: Intensive Group — Participants in this group would receive print materials on diet and exercise and attend group sessions that would meet weekly for the first 4 months, then every two weeks for the next 2 months, and then monthly for the next 6 months over the course of one year.
  Arms: Intensive Group

SUMMARY:
The purpose of the ENERGY trial is to explore whether two different programs that are focused on weight management, through increased exercise and a healthy diet, are feasible, and have an impact on body weight, quality of life and fatigue. Since obesity among breast cancer survivors is associated with recurrence and other co-morbidities, those will be assessed and their impact calculated. Blood samples will be collected to enable analysis of potential mechanisms and differential response across subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer (stages I (≥1 cm), stage II, or stage IIIA, B, C excluding distant metastasis) diagnosed between 6 months and 5 years earlier; after initial therapies are completed, diagnosed between six months and five years earlier
* BMI between 25 to 45 kg/m2
* Able to comply with all required study procedures and schedule

Exclusion Criteria:

* Serious medical condition or psychiatric illness
* Inability to be moderately physically active
* Obesity of known endocrine origin (e.g., untreated hypothyroidism, PCOS)
* Currently enrolled in a weight loss program
* Current use of weight loss medication or supplements
* Previous surgical procedures for weight reduction
* Planning weight loss surgery in the next 2 years.
* 6+ months use of meds likely to cause weight gain or prevent weight loss
* Planned surgical procedure that can impact the conduct of the study
* Currently pregnant/breastfeeding
* Planning to become pregnant within the next 2 years
* Have plans to relocate from area within 2 years
* Family relative or close friend is a trial staff member or a study participant
* Any condition which in the opinion of the investigator makes the subject unsuitable for inclusion in this study

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2010-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Weight loss | 2 years

SECONDARY OUTCOMES:
Improvement in quality of life | 2 years
Improvement in fatigue | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl L. Rock, PhD, RD, Principal Investigator — University of California, San Diego
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Moores UCSD Cancer Center, La Jolla, California
  - University of Colorado Denver, Aurora, Colorado
  - Washington University in St. Louis:, St Louis, Missouri

REFERENCES:
- [Derived] Kenzik KM, Demark-Wahnefried W, Ganz PA, Colditz G, Rock CL, Rogers LQ. Changes in Body Mass Index and Physical Activity Predict Changes in Vitality During a Weight Loss Trial in Breast Cancer Survivors. Ann Behav Med. 2018 Nov 12;52(12):999-1009. doi: 10.1093/abm/kay004. PMID 29617707
- [Derived] Rock CL, Flatt SW, Byers TE, Colditz GA, Demark-Wahnefried W, Ganz PA, Wolin KY, Elias A, Krontiras H, Liu J, Naughton M, Pakiz B, Parker BA, Sedjo RL, Wyatt H. Results of the Exercise and Nutrition to Enhance Recovery and Good Health for You (ENERGY) Trial: A Behavioral Weight Loss Intervention in Overweight or Obese Breast Cancer Survivors. J Clin Oncol. 2015 Oct 1;33(28):3169-76. doi: 10.1200/JCO.2015.61.1095. Epub 2015 Aug 17. PMID 26282657